CLINICAL TRIAL: NCT07201740
Title: The Effectiveness of Leap Motion-Based Virtual Reality in the Rehabilitation of Flexor Tendon Injuries of the Hand
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Serkan Kablanoğlu, PhD, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KC-KABLANOGLU-001
Record Dates: First submitted 2025-08-26; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-08

CONDITIONS: Flexor Tendon Injuries of the Hand (Zones II-V)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Arm Title: Leap Motion + Routine Hand Rehabilitation
  Description: Participants receive standard postoperative hand rehabilitation plus Leap Motion-based virtual reality training for 20 minutes/day, 5 days/week, for 4 weeks.
  Intervention Type: Device (Leap Motion-based virtual reality therapy)
  Other Intervention: Behavioral (Routine hand rehabilitation program)
  Interventions: Device: Leap Motion-based Virtual Reality Therapy
- Active Comparator (Control) (Active Comparator): Arm 2 - Active Comparator (Control)
  Arm Title: Routine Hand Rehabilitation Only
  Description: Participants receive only routine postoperative hand rehabilitation for 1 hour/day, 5 days/week, for 4 weeks.
  Intervention Type: Behavioral (Routine hand rehabilitation program)
  Interventions: Other: Active Comparator - Routine Rehabilitation Only

INTERVENTIONS:
Device: Leap Motion-based Virtual Reality Therapy — Arm 1 - Experimental (Leap Motion + Routine Hand Rehabilitation)
  Intervention Description: Participants will receive standard postoperative hand rehabilitation plus Leap Motion-based virtual reality training. The VR training will be performed for 20 minutes per day, 5 days per week, for 4 weeks, in addition to routine rehabilitation. The Leap Motion Controller tracks hand and finger movements without physical contact and allows participants to practice functional tasks and grasp patterns in a virtual environment.
  Arm 2 - Active Comparator (Routine Hand Rehabilitation Only)
  Intervention Description: Participants will receive only routine postoperative hand rehabilitation, performed for 1 hour per day, 5 days per week, for 4 weeks, supervised by a therapist.
  Arms: Experimental
Other: Active Comparator - Routine Rehabilitation Only — Participants will receive only routine postoperative hand rehabilitation, performed for 1 hour per day, 5 days per week, for 4 weeks, supervised by a therapist.
  Arms: Active Comparator (Control)

SUMMARY:
This randomized controlled clinical trial aims to evaluate the effectiveness of a Leap Motion-based virtual reality rehabilitation program in patients who underwent surgical repair for flexor tendon injuries of the hand (zones II-V). A total of 66 participants, aged 18-65 years and at least 5 weeks postoperative, will be randomly assigned to two groups: the intervention group will receive routine hand rehabilitation plus Leap Motion-based virtual reality therapy for 20 minutes per day, 5 days per week, for 4 weeks; while the control group will continue routine hand rehabilitation only. Outcomes will include joint range of motion measured with a goniometer, pain intensity assessed with a Visual Analog Scale (VAS), grip strength measured with a Jamar dynamometer, and functional outcomes assessed using the QuickDASH questionnaire. The primary endpoint is the change in range of motion, grip strength, and QuickDASH score from baseline to post-treatment. Secondary endpoints include changes in upper extremity function and pain tolerance. All interventions will be delivered under therapist supervision. This study is expected to provide evidence on whether integrating Leap Motion-based virtual reality into conventional rehabilitation improves clinical outcomes after flexor tendon repair.

ELIGIBILITY:
Inclusion Criteria:

Age between 18 and 65 years

Flexor tendon injury of the hand (zones II-V)

Early surgical repair completed

At least 5 weeks postoperative

Eligible for routine hand rehabilitation program

Exclusion Criteria:

Communication problems

Cognitive impairment

Additional musculoskeletal, neurological, or rheumatological diseases affecting upper extremity function

Multiple trauma cases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Upper limb disability/function | Baseline and 4 weeks post-treatment
  Functional disability of the upper limb assessed with the Quick Disabilities of the Arm, Shoulder, and Hand questionnaire. In the Q-DASH, a higher score indicates worse outcome, while a lower score indicates better outcome.
Joint range of motion (ROM) | Baseline and 4 weeks post-treatment
  Assessed with a manual goniometer. Comparison between baseline and after 4 weeks of treatment. A higher ROM indicates a better clinical condition.
Grip strength | Baseline and 4 weeks post-treatment
  Assessed using a Jamar hand dynamometer.